CLINICAL TRIAL: NCT04862598
Title: Virtual Reality to Improve Satisfaction in Patients Undergoing Hysteroscopy: A Single-centre Randomized Controlled Trial
Brief Title: Virtual Reality to Improve Satisfaction in Hysteroscopy Patients
Acronym: VIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Anthony Chau, Clinical assistant professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H20-03663
Record Dates: First submitted 2021-02-23; First posted 2021-04-28 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Patient Satisfaction; Virtual Reality; Hysteroscopy
Keywords: Virtual Reality; Hysteroscopy; Iowa Satisfaction Scale; Sedation
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The patient will be positioned on the operating table and have routine monitoring attached (ECG, blood pressure, O2 saturations, end tidal carbon dioxide monitoring (ETCO2). A surgical safety time out will be performed. The patient will receive routine operative and nursing care. The study team member will record highest and lowest heart rate and blood pressure as well as lowest O2 saturation and the total intra-operative dose of fentanyl and midazolam administered to the patient. At the end of the procedure, the patient is assisted into a wheelchair and will return to the recovery area. After 15 minutes of recovery, a member of the study team will give them the post-operative questionnaires which will consist of answering how anxious they felt during the procedure and the 11 question Iowa Satisfaction with Anesthesia scale (ISAS). The patient will then be free to leave once they have met the standard discharge criteria.
- VR Group (Experimental): The patient wears the VR headset after being positioned on the table and the surgical time out has been completed. The VR scene and accompanying music will continue until the end of the procedure or until the patient wishes for it to be removed. The patient will receive standard operative and nursing care. The study team member will record the intra-operative vitals as detailed in the control group procedure. At the end of the procedure, the patient will be moved to recovery and will receive standard care. At 15 minutes, they will be provided with the anxiety questionnaire and the ISAS. Additional questions will be asked; their level of VR immersion and if they would like to receive the VR technology again if they were to undergo another procedure in the future. They will then be free to leave once they have met the standard discharge criteria.
  Interventions: Device: Oculus Virtual Reality

INTERVENTIONS:
Device: Oculus Virtual Reality — The patient will receive standard care, augmented with virtual reality. Their post-operative satisfaction score will be recorded.
  Arms: VR Group

SUMMARY:
This study aims to investigate whether viewing an immersive virtual reality (VR) image through a VR headset during elective hysteroscopy under Registered Nurse (RN) led sedation with fentanyl and midazolam plus local anesthesia (monitored anesthetic care) will improve patient satisfaction with their anesthesia. Patients will be randomized to either receive usual care or usual care plus VR. Satisfaction will be measured by asking patients to complete a post-procedure survey consisting of 11 questions.

DETAILED DESCRIPTION:
Purpose: To determine whether viewing an immersive VR image (viewed over an Oculus Quest VR headset) during hysteroscopy can improve patient satisfaction with their anesthesia (sedation plus local anesthesia). The VR image used in the study is Cosmic Flow: A Relaxing VR experience, which is freely available from Oculus. The patient will also wear headphones during the study which will play relaxing meditation music.

Hypothesis: The use of immersive VR during elective hysteroscopy under sedation will improve patient satisfaction with their anesthesia by at least 20%, measured using the Iowa Satisfaction with Anesthesia Scale.

Justification: Ambulatory hysteroscopy is conducted under general anesthesia or in the established Procedural Sedation Program. The latter involves Registered Nurse (RN) led sedation, consisting of the administration of sedation (midazolam) and analgesia (fentanyl) to reduce discomfort and anxiety. However, these medications have unwanted side-effects such as over-sedation and nausea, which can delay discharge and reduce patient satisfaction with their procedure. To minimize these complications, non-pharmacological therapy is of interest, as it aims to reduce the need and dosage of these medications. Virtual reality is one such non-pharmacological intervention which has been trialled in several settings, and has been shown to have beneficial effects on pain and anxiety during procedures such as wound dressing changes, upper GI endoscopies and dental procedures. Virtual reality use in the healthcare setting is currently in an early phase of research, and more study is needed on effects of VR on precise outcomes such as patient satisfaction, which is an important marker for quality in healthcare.

Objectives: The objective is to study patient reported satisfaction with their anesthesia (sedation plus local anesthesia) when they receive standard care to when they receive standard care plus viewing an immersive VR image during their hysteroscopy procedure.

Research Design: This is a randomized controlled trial involving data collection before, during and after the hysteroscopy procedure.

Statistical Analysis: The primary outcome in change in patient satisfaction scores will be compared using paired t-test. For secondary outcomes, all continuous data will be compared using t-test or Mann-Whitney U test as appropriate. Incidence and proportion outcomes will be analyzed using Fisher exact test.

ELIGIBILITY:
Inclusion Criteria:

* Indications for hysteroscopy under RN-provided sedation

Exclusion Criteria:

* Inability to provide informed consent to participate in the study (e.g. significant language barrier)
* Severe cognitive impairment
* Chronic benzodiazepine use
* Chronic opioid use
* Presence or history of psychotic psychiatric disorders
* Presence or history of seizure disorders
* Visual acuity <1 with correction
* Hearing impairment requiring correction

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 15 minutes post-operatively
  Change in post-procedure patient satisfaction score (Iowa Satisfaction Scale) of at least 0.6 between the Virtual Reality group and the control group. High scores are better than low scores which are worse. Scores range from -3 (completely unsatisfied) to 3 (completely satisfied)

SECONDARY OUTCOMES:
Patient anxiety scores before and after the procedure | 30 minutes before operation (one anxiety score). 15 minutes after operation (one anxiety score). On a 10 point Likert anxiety scale (0-10) high scores are more anxious and low scores are less anxious.
  10-point Likert Scale
Total Fentanyl dose | 45 minutes throughout the operation
  Total IV Fentanyl dose in mcgs during the procedure
Total Midazolam dose | 45 minutes throughout the operation
  Total IV Midazolam dose in mgs during the procedure
Occurrence of intraoperative hemodynamic changes | 45 minutes throughout the operation
  Increase/decrease of 30 percent of SBP or HR compared to baseline
Incidence of desaturation | 45 minutes throughout the operation
  Pulse oxygen saturation <90 percent
Incidence of early termination of VR experience | Noted during the procedure
  Noting whether the patient decides to terminate the VR experience before the end of their procedure.
Proportion of patients wishing to use the technology again | Noted 15 minutes after the operation
  Yes/No response
Immersion perception score of the VR system | 15 minutes after the operation.
  10 point Likert scale. On a 10 point Likert immersion scale (0-10) high scores are more immersed and low scores are less immersed.

OTHER OUTCOMES:
Reason for early termination of VR experience | 45 minutes throughout the operation
  Reasons may include: Patient desire/Medical decision/Nausea/Vomiting/Dizziness/ Headache/Device failure/ other

CONTACTS AND LOCATIONS:
Overall Officials: Anton Chau, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada